CLINICAL TRIAL: NCT04570527
Title: Effects and Mechanism of Adipokines Cardiac Protection in Obese Patients With Coronary Artery Disease (CAD)
Brief Title: Optimized Cardioprotection Therapy in Obese Subjects With CAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, sunddong, Cardiology department, Xijing Hospital
Other Study IDs: OB-CAD
Record Dates: First submitted 2020-09-25; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Coronary Artery Disease (CAD) (E.G., Angina, Myocardial Infarction, and Atherosclerotic Heart Disease (ASHD)); Obesity; Adiposis; Heart
Keywords: Coronary artery disease; Adipokines; Obesity; Diabetes mellitus
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Myocardial Infarction; Obesity; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Serum, Plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obesity: BMI>=25
  Interventions: Procedure: PCI
- Non-Obesity: BMI<25
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI — percutaneous coronary intervention

SUMMARY:
The purpose of this study is to investigate the efficacy and mechanism of Adipokines Cardiac Protection in Obese Patients With coronary artery disease (CAD).

DETAILED DESCRIPTION:
Adipokines (or adipocytokines) can be defined as a group of more than 600 bioactive molecules made from adipose tissue that acts as paracrine and endocrine hormones. Adipokines are involved in maintaining varieties of processes such as, appetite and satiety, energy expenditure activity, endothelial function, blood pressure, hemostasis, adipogenesis, insulin sensitivity, energy metabolism in insulin-sensitive tissues, fat distribution and insulin secretion in pancreatic β-cells. Adipokines may contribute to reduce scar formation and improve cardiac function in coronary artery disease (CAD). Reperfusion therapy such as percutaneous coronary intervention (PCI) should be administered to all eligible patients with CAD symptom. However, our previous work showed that obese patients may benefit more from PCI. Thus, the aim of the present study was to investigate the efficacy and mechanism of adipokines cardiac protection for obese and non-obese patients with coronary artery disease (CAD).

ELIGIBILITY:
Inclusion Criteria:

coronary artery disease according to the WHO definition With or without percutaneous coronary intervention

Exclusion Criteria:

previous Coronary artery bypass grafting (CABG) cardiomyopathy atrial fibrillation or flutter previous heart surgery severe valvular heart disease disease of the hematopoietic system NYHA functional class IV heart failure at baseline severe renal, lung and liver disease cancer

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of CAD were enrolled in this study
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of patient death during the follow up period | 1 year

SECONDARY OUTCOMES:
Left ventricular ejection fraction | 1 year
Number of target vessel revascularization | 1 year
Angina class according to the canadian cardiovascular society (CCS) classification | 1 year
Scores on the Seattle angina questionnaire | 1 year
six-min walk distance (6MWD) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dongdong Sun, MD, PhD, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Zhang X, Duan Y, Zhang X, Jiang M, Man W, Zhang Y, Wu D, Zhang J, Song X, Li C, Lin J, Sun D. Adipsin alleviates cardiac microvascular injury in diabetic cardiomyopathy through Csk-dependent signaling mechanism. BMC Med. 2023 May 26;21(1):197. doi: 10.1186/s12916-023-02887-7. PMID 37237266